CLINICAL TRIAL: NCT02948699
Title: A Prospective, Randomized Controlled Open Research About the Impact of Nutritional Support on the Radiation Tolerance and Clinical Outcomes for Local Advanced Nasopharyngeal Carcinoma Patients
Brief Title: A Research About Nutrition Impact for Local Advanced Nasopharyngeal Carcinoma Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NPC-NUTR-2016
Record Dates: First submitted 2016-10-21; First posted 2016-10-28 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Malignant Neoplasm of Nasopharynx
Keywords: nasopharyngeal carcinoma; intensity-modulated radiotherapy; nutrition support; nutrition assessment
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrition support (Experimental): Nutrison was added to regular diet while the patients can be fed through mouth. Nutrison will replace regular diet by NG or PEG while the patients can not eat for serious oral mucositis.
  Interventions: Dietary Supplement: Nutrison
- Regular diet (No Intervention): Regular diet without other nutritional intervention.

INTERVENTIONS:
Dietary Supplement: Nutrison — Nutrison(400-600ml/d) will be given to Arm 1 patient between regular diet. When the daily ration was cut down to 50%,100ml/h Nutrison was added. When grade Ⅲ-Ⅳ oral mucositis appeared, total Nutrison was applied to patients by NG or PEG.
  Arms: Nutrition support

SUMMARY:
The chemo-radiotherapy for the local advanced nasopharyngeal carcinoma patients will induce the mucosal ulcer and damage salivary glands. Consequently, it can disturb the nutrition conditions and clinical outcomes of patients. This research tries to evaluate the nutrition status at the baseline, before and after radiotherapy, during the follow-up by the body mass index, hematological indexes, immunological indexes, and nutrition questionnaires including PG-SGA and NRS 2002. Through the evaluation of two different nutritional interventions, the investigators aim to find an optimized assessment model and the best nutrition support patterns.

DETAILED DESCRIPTION:
All nasopharyngeal patients received radical treatment including neo-adjuvant chemotherapy and concurrent chemo-radiotherapy. At the beginning, the investigators assign patient to experimental and control groups randomly. Patients in experimental group received standard nutritional support by adding NUTRISON. Control patients will give conventional nutritional guidance. The investigators collected all the nutritional indexed at first visit, before and after radiotherapy, 1, 3, 6, 9, 12 months after radiotherapy. All these data will be set into statistical software to produce an optimized model for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically conformed Initial nasopharyngeal carcinoma
2. Patients can feed through the mouth.
3. ECOG (Eastern Cooperative Oncology Group) : 0-2.
4. No history of chemo-radiotherapy, immuno-therapy or biotherapy.
5. Normal hemodynamic indices before the recruitment (including white blood cell count>4.0×109/L, neutrophil count>1.5×109/L, platelet count >100×109/L, hemoglobin≥90g/l, normal liver/kidney function).
6. Informed consent signed.

Exclusion Criteria:

1. History of malignant tumors.
2. Any severe complications contraindicated chemotherapy or radiotherapy.
3. Medical history of central nervous system, cognitive or psychological diseases;
4. Pregnant or nursing women.
5. Patients with mental disease cannot complete the questionaire.
6. Patients refused the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  From the first treatment to the death of any causes

SECONDARY OUTCOMES:
Progress free survival | 5 years
  From the first treatment to the progress of diseases

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhejiang Cancer Hosptial, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No